CLINICAL TRIAL: NCT02302625
Title: Exposure-based CBT for Itching in Atopic Dermatitis
Brief Title: Cognitive Behavior Therapy for Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Hedman, Phd, psychologist, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBT atopic
Record Dates: First submitted 2014-11-19; First posted 2014-11-27 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Atopic Dermatitis
Keywords: Cognitive behavior therapy
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive behavior therapy (Experimental): Cognitive behavior therapy based on exposure and response prevention. The treatment also incorporates mindfulness training as a means to increasing tolerance for aversive thoughts and emotions associated with AD. The treatment is delivered by a licensed psychologist and comprises 10 individual weekly sessions.
  Interventions: Behavioral: Cognitive behavior therapy

INTERVENTIONS:
Behavioral: Cognitive behavior therapy — Cognitive behavior therapy based on exposure and response prevention. The treatment also incorporates mindfulness training as a means to increasing tolerance for aversive thoughts and emotions associated with AD. The treatment is delivered by a licensed psychologist and comprises 10 individual weekly sessions.

SUMMARY:
Atopic dermatitis is an inflammatory skin disease characterized by itching, dry skin and recurrent inflammatory eczema. It is one of the most common skin diseases and is associated with reduced quality of life, functional impairment and sleep difficulties. The present study aims to investigate a new exposure-based cognitive behavioral psychological treatment for the disorder. The trial is a small scale open trial (n=25) with assessments at baseline, post-treatment and 6-month follow-up. The primary outcome is the SCORAD.

DETAILED DESCRIPTION:
Atopic dermatitis (AD)is an inflammatory skin disease characterized by itching, dry skin and recurrent inflammatory eczema. It is one of the most common skin diseases and is associated with reduced quality of life, functional impairment and sleep difficulties. There are currently no pharmacological treatments that are effective in curing the disorder in the longer-term. Itching is one of the core symptoms in AD and it has been shown that the behavioral response to itching, scratching, has a maintaining function in AD. Reducing scratching may therefore play an important role in alleviating AD. Although behavioral aspects play a significant role in AD only a few studies have investigated the effect of psychological treatment for AD. These studies have shown promising results and the present study aim to add to the body of knowledge by testing a new form of cognitive behavioral treatment for AD. This new treatment is based on the idea that patients could benefit from training in exposure to events that could lead to increase in itching while refraining from scratching. To enable this the treatment incorporates more recently developed cognitive behavioral components such as mindfulness training.

The present study aims to investigate a new exposure-based cognitive behavioral psychological treatment for the disorder. The trial is a small scale open trial (n=25) with assessments at baseline, post-treatment and 6-month follow-up. The primary outcome is the SCORAD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD with at least moderate severity
* AD for at least 6 months
* Age 18-65
* Ability to read and write in Swedish

Exclusion Criteria:

* Serious psychiatric illness
* Concurrent light treatment or peroral treatment for AD
* Pregnancy
* Other concurrent or recently finished psychological treatment for AD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Severity Scoring of Atopic Dermatitis index (SCORAD) | Change from baseline to 10 weeks follow-up and 6-month follow-up

SECONDARY OUTCOMES:
Beck Anxiety Inventory | Change from baseline to 10 weeks follow-up and 6-month follow-up
Montgomery-Åsberg Depression Rating Scale-Self-rated | Change from baseline to 10 weeks follow-up and 6-month follow-up
Quality of Life Inventory | Change from baseline to 10 weeks follow-up and 6-month follow-up
Alcohol Disorders Identification Test | Baseline only
SRH-5 | Change from baseline to 10 weeks follow-up and 6-month follow-up
Trimbos and Institute of Technology Cost Questionnaire for Psychiatric illness (TIC-P) | Change from baseline to 10 weeks follow-up and 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Erik Hedman, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet and Gustavsberg primary care center, Stockholm, Stockholm County, Sweden